CLINICAL TRIAL: NCT03970343
Title: A Prospective, Multi-center, Non-randomized, Single Arm Open Label Study of 620 Subjects Receiving the OPTIMIZER Smart With CCM Therapy as Standard of Care
Brief Title: Post Approval Study (PAS) of the OPTIMIZER Smart and CCM Therapy
Acronym: PAS
Status: Active, not recruiting | Type: Observational
Sponsor: Impulse Dynamics (Industry)
Responsible Party: Sponsor
Other Study IDs: CA_CP_307
Record Dates: First submitted 2019-05-23; First posted 2019-05-31 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-11

CONDITIONS: Heart Failure
Keywords: OPTIMIZER; Heart Failure; CCM; Post-Approval Study; NYHA class III; FIX-HF-5C; Chronic heart failure; Ejection fraction between 25 and 45; cardiac contractility modulation
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

INTERVENTIONS:
Device: OPTIMIZER Smart System — Eligible subjects will receive the OPTIMIZER Smart, which is comprised of three major components:
  1. Optimizer Smart or Optimizer Smart Mini
  2. Vesta Charger or Guardio Charger
  3. Two commercially available intravascular leads

SUMMARY:
The OPTIMIZER Smart Post-Approval Study is a prospective, multi-center, non-randomized, single arm open label study of 620 subjects receiving an OPTIMIZER implant as standard of care. Patients to be included will have NYHA functional class III symptoms and a left ventricular ejection fraction of 25-45%

DETAILED DESCRIPTION:
The Impulse Dynamics OPTIMIZER Smart Pre-Market Application (PMA) clinical data confirmed that CCM therapy delivered with the Optimizer meaningfully improved health outcomes in patients with NYHA class III heart failure symptoms and left ventricular ejection fraction of 25-45%. CCM has shown significant improvements in quality of life measures, with an average improvement of >11 points in MLHWFQ incremental to the improvement of a randomized control group with no device. Six minute hall walk and functional class also showed improvements in the PMA data. The post-approval study (PAS) protocol has been designed to evaluate long term safety and efficacy of the OPTIMIZER Smart in a real-world setting.

ELIGIBILITY:
Inclusion Criteria:

1. Patient provides written authorization and/or consent per institution and geographical requirements
2. Male or non-pregnant female, aged 18 or older
3. Left ventricular ejection fraction of 25-45% (inclusive, per site assessment)
4. NYHA Class III heart failure symptoms
5. Stated willingness to comply with all study procedures and availability for the duration of the study
6. Patient has been treated with guideline-directed medical therapy

Exclusion Criteria:

1. Primary heart failure due to uncorrected mitral valve disease, or mitral valve repair or clip within 90 days of implant
2. IV inotropes, hemofiltration, or any form of positive inotropic support within 30 days prior to implant
3. Myocardial infarction within 90 days prior to implant
4. Undergone a CABG procedure within 90 days or a PTCA procedure within 30 days of implant
5. Prior heart transplant or ventricular assist device
6. Mechanical tricuspid valve
7. Receiving cardiac resynchronization therapy (CRT) or has a Class I indication for CRT implantation according to the ACCF/AHA/HRS guidelines for device-based therapy
8. Participating in a cardiac investigational study at the same time
9. Patient is in a vulnerable population (such as significant mental disability, prisoner) that in the judgement of the PI impedes ability to provide informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants will represent a patient population with stable, systolic left ventricular dysfunction and moderate symptomatic heart failure despite guideline-directed medical therapy.
Sampling Method: Probability Sample
Enrollment: 620 (Estimated)
Dates: Start 2020-01-21 (Actual); Primary Completion 2028-07 (Estimated); Study Completion 2028-07 (Estimated)

PRIMARY OUTCOMES:
Incidence of procedure and device-related complications | 1 year
  Demonstrate, in the post-approval setting, that the OPTIMIZER Smart is safe to use, by assessing the rate of procedure related complications (30 days) and device related complications (1-year)
All-cause mortality | 3 years
  Observed mortality will be compared to the predicted mortality according to the Seattle Heart Failure Model (SHFM) at 1 year and 3 years post-implant
Procedure related complications | 30-days
  Procedure related complications through the end of 30 days following the index procedure

SECONDARY OUTCOMES:
Cardiovascular hospitalizations | 2 years
  Change in cardiovascular hospitalization rate and HF hospitalization rate from 1-year prior to 2 years following index implantation

CONTACTS AND LOCATIONS:
Overall Officials: Rami Kahwash, MD, Study Director — Ohio State University; Raul Weiss, MD, Study Director — Mt. Sinai Miami
Locations (90):
- United States (90):
  - CardioVascular Associates of Mesa (CVAM), Mesa, Arizona
  - Chan Heart Rhythm Institute (CHRI), Mesa, Arizona
  - Southwest Cardiovascular Associates, Mesa, Arizona
  - Banner University Medical Center, Phoenix, Arizona
  - Cardiovascular Society of Arizona, Phoenix, Arizona
  - Arizona Cardiovascular Research Center, Phoenix, Arizona
  - Honor Health, Scottsdale, Arizona
  - Pima Heart and Vascular Research Center, Tucson, Arizona
  - University of AZ - Sarver Heart Center, Tucson, Arizona
  - Cardiovascular Institute of San Diego, Chula Vista, California
  - NorthBay Health, Heart and Vascular, Fairfield, California
  - Mid Valley Cardiology - Fresno, Fresno, California
  - South Orange County Cardiology Group, Laguna Hills, California
  - University of Southern California - Keck School of Medicine, Los Angeles, California
  - Cedars-Sinai Medical Center, Los Angeles, California
  - Valley Clinical Trials, Northridge, California
  - Valley Clinical Trials, Pasadena, California
  - Torrance Memorial Medical Center, Torrance, California
  - Aurora Denver Cardiology Associates, Aurora, Colorado
  - MedStar Washington Hospital Center, Washington D.C., District of Columbia
  - Heart Rhythm Solutions, Davie, Florida
  - Florida Memorial Hospital, Jacksonville, Florida
  - Florida Cardiology, Orlando, Florida
  - Florida Heart Rhythm Specialist, Plantation, Florida
  - Piedmont Heart, Atlanta, Georgia
  - Redmond Regional Medical Center, Rome, Georgia
  - Advocate Illinois Masonic Medical Center, Chicago, Illinois
  - Advocate Good Samaritan Hospital, Downers Grove, Illinois
  - OSF Healthcare Cardiovascular Institute, Peoria, Illinois
  - OSF HealthCare Cardiovascular Institute, Rockford, Illinois
  - OSF Healthcare Cardiovascular Institute, Urbana, Illinois
  - Franciscan Physician Network, Indianapolis, Indiana
  - Ascension St. Vincent, Indianapolis, Indiana
  - Community Healthcare System, Munster, Indiana
  - Baptist Lexington, Lexington, Kentucky
  - University of Kentucky - Gill Heart & Vascular Institute Clinical Research, Lexington, Kentucky
  - Massachusetts General Hospital, Boston, Massachusetts
  - Ascension Providence Park Hospital, Novi, Michigan
  - St. Joseph Mercy Oakland, Pontiac, Michigan
  - Downriver Heart and Vascular, Southgate, Michigan
  - Trinity Health Michigan Heart, Ypsilanti, Michigan
  - Minneapolis Heart Institute Foundation - Allina, Minneapolis, Minnesota
  - St. Louis Heart and Vascular, Bridgeton, Missouri
  - Logan Health, Kalispell, Montana
  - Cooper Hospital, Haddon Heights, New Jersey
  - Virtua Health - Our Lady of Lourdes, Marlton, New Jersey
  - Morristown Medical Center, Morristown, New Jersey
  - Rutgers Medical School, Newark, New Jersey
  - Valley Hospital, Ridgewood, New Jersey
  - Mount Sinai Morningside, New York, New York
  - Mission Health, Asheville, North Carolina
  - Atrium Health, Charlotte, North Carolina
  - NC Heart and Vascular Research, Raleigh, North Carolina
  - TriHealth Hatton, Cincinnati, Ohio
  - University Hospitals of Cleveland Medical Center, Cleveland, Ohio
  - The Ohio State University, Columbus, Ohio
  - Mount Carmel Research institute, Columbus, Ohio
  - Regional Cardiac Arrythmia Inc., Steubenville, Ohio
  - ProMedica Health Systems, Toledo, Ohio
  - Mercy Health - St. Vincent Medical Center, Toledo, Ohio
  - Oklahoma Heart Hospital, Oklahoma City, Oklahoma
  - St. Luke's University Health Network, Allentown, Pennsylvania
  - Bryn Mawr Hospital, Bryn Mawr, Pennsylvania
  - UPMC Pinnacle Health, Harrisburg, Pennsylvania
  - Penn State Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - Penn Medicine Lancaster General Hospital, Lancaster, Pennsylvania
  - Cardiology Consultants of Philadelphia, Philadelphia, Pennsylvania
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - Penn Presybyterian Medical Center, Philadelphia, Pennsylvania
  - Temple University Hospital, Philadelphia, Pennsylvania
  - Einstein Medical Center, Philadelphia, Pennsylvania
  - Allegheny General Hospital, Pittsburgh, Pennsylvania
  - UPMC Heart and Vascular Institute, Pittsburgh, Pennsylvania
  - Reading Hospital, Reading, Pennsylvania
  - Cardiovascular Consultants of Philadelphia, Yardley, Pennsylvania
  - Texas Cardiac Arrhythmia Research, Austin, Texas
  - VA North Texas Medical Center, Dallas, Texas
  - Texan Procedure Center, El Paso, Texas
  - Baylor College of Medicine, Houston, Texas
  - UT Health - Memorial Hermann Hospital, Houston, Texas
  - Heart and Rhythm Institute of South Texas, San Antonio, Texas
  - UT Health San Antonio, San Antonio, Texas
  - CHRISTUS Trinity Clinic Research, Tyler, Texas
  - Centra Health- Lynchburg General Hospital, Lynchburg, Virginia
  - Bon Secours St. Mary's Hospital, Midlothian, Virginia
  - HCA Chippenham Hospital, Richmond, Virginia
  - Richmond VA Medical Center, Richmond, Virginia
  - CAMC Clinical Trials Center, Charleston, West Virginia
  - Marshall Cardiology, Huntington, West Virginia
  - Aurora Research Institute, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: No